CLINICAL TRIAL: NCT06485076
Title: Phase II Feasibility Study of Early Palliative Care for Patients With Multiple Myeloma and Aggressive Lymphoma
Brief Title: Early Palliative Care for Patients With Multiple Myeloma and Aggressive Lymphoma
Acronym: EPC-MM+L
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Myeloma Canada (Unknown); The Leukemia and Lymphoma Society of Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DeGasperis
Record Dates: First submitted 2024-03-25; First posted 2024-07-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory; Multiple Myeloma Stage III; Multiple Myeloma Progression; Multiple Myeloma; B Cell Lymphoma; Lymphoma, B-Cell; Aggressive Lymphoma
Keywords: early palliative care; multiple myeloma; quality of life; symptom management; aggressive lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, B-Cell

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Palliative Care (Experimental): Patients in the intervention/early palliative care arm will be invited to attend a consultation (in-person or via Microsoft Teams) in the outpatient palliative care clinic alongside ongoing care from their hematologist. The intervention will comprise of a comprehensive interdisciplinary assessment from a specialist palliative care nurse and a physician within two weeks of referral and monthly follow-up visits (in-person, via Microsoft Teams, or via phone) for 3 months. This will include an assessment of physical symptoms, psychological distress, social supports and advance care planning, as well as 24/7 telephone support between visits, community-based resources, and access to the acute palliative care unit, if required. Caregivers of these patients will be encouraged to attend at least one palliative care clinic visit with the patient.
  Interventions: Other: Early Palliative Care
- Usual Care (No Intervention): Patients in the usual care arm will receive care from their hematologist as usual, with referral to the outpatient palliative care clinic at the discretion of the hematologist or upon patient request

INTERVENTIONS:
Other: Early Palliative Care — see previous description
  Arms: Early Palliative Care

SUMMARY:
Patients with multiple myeloma experience a wide range of physical and psychological symptoms from the time of their diagnosis. Meanwhile, patients with aggressive lymphomas undergo unpredictable illness courses, resulting in goals of care conversations occurring late in the illness trajectory and aggressive care being received in the last 30 days of life. Early palliative care alongside usual cancer care has been shown to improve patient outcomes such as symptom burden, mood, and quality of life in patients with solid tumours (e.g. lung, breast or gynecological cancers), but has not been explored among patients with blood cancers to date.

The goal of this clinical trial is to a brief early palliative care intervention for patients with multiple myeloma and aggressive B cell lymphoma and their caregivers (lymphoma only) attending the Princess Margaret Cancer Centre. The main goals of the study are:

* To see if it is possible to apply the early palliative care intervention for patients with multiple myeloma and aggressive lymphoma and their caregivers (lymphoma only)
* To see if this early palliative care intervention works well for these patients and caregivers
* To compare patient and caregiver experiences with early palliative care and usual care
* To explore perceptions and experiences of providing palliative care among healthcare providers involved in the care of these patients and caregivers.

Patients, and their respective caregivers if participating, will be randomly assigned to one of two groups: one group will receive early palliative care in addition to usual care from their blood cancer doctor, and the other group will receive usual care from their blood cancer doctor only. All participants will be asked to fill out questionnaires about their quality of life, symptom burden, mood, and satisfaction with care throughout the study. Researchers will compare the results between the two groups to see if there are any improvements in quality of life for the patients who received early palliative care and their caregivers.

Some patients and caregivers will be asked to take part in interviews at the end of the trial to answer questions about their experience taking part in the study. Some healthcare providers who care for these patients will also be asked to take part in interviews at the end of the trial to describe their perceptions and experiences of providing palliative care.

The researchers will use the results of this study to guide in the development of a larger clinical trial.

DETAILED DESCRIPTION:
In this study, the investigators will test an early palliative care intervention for patients with multiple myeloma and aggressive B cell lymphoma and their caregivers (lymphoma only) in a randomized phase II trial in which outpatients and their caregivers will be allocated to one of two groups: symptom screening alone (usual care) or early palliative care alongside usual care (intervention).

Participants will be recruited from multiple myeloma and lymphoma outpatient clinics at the Princess Margaret Cancer Centre. Consenting patients and caregivers will complete questionnaires measuring outcomes of quality of life, symptom burden, depression, and satisfaction with care at recruitment, 1 month, 2 months, and 3 months. After the 3-month follow-up time point, select patients and caregivers will complete a one-time semi-structured interview that explores their experiences taking part in the study. Select healthcare providers from the multiple myeloma, lymphoma, and palliative care teams will also be invited to participate in a one-time focus group or individual interview. Healthcare providers in malignant hematology will be asked to describe their perceptions of palliative care and providers in palliative care will be asked to describe their experiences providing palliative care to patients with multiple myeloma and aggressive lymphoma and their caregivers.

The purposes of this phase II trial are to:

1. Assess the feasibility of early palliative care for outpatients with multiple myeloma and aggressive lymphoma and their caregivers (lymphoma only).
2. Assess preliminary efficacy of early palliative care for these outpatients and caregivers.
3. Qualitatively compare patient and caregiver experiences and perceptions of palliative care between the intervention and usual care arms of the study.
4. Qualitatively describe perceptions of palliative care among healthcare providers in malignant hematology, as well as the experiences of providing palliative care to patients with multiple myeloma and aggressive lymphoma among healthcare providers in palliative care.

Feasibility criteria are: (i) accrual of at least 80 patients (40 with multiple myeloma and 40 with aggressive B cell lymphoma) and up to 40 caregivers of patients with aggressive B cell lymphoma over 12 months; (ii) ≥60% of recruited patients and caregivers complete self-reported outcomes (PROs) at baseline, and monthly for three months; and (iii) ≥60% of patients and their caregivers in the intervention arm have at least one visit to the palliative care clinic.

ELIGIBILITY:
Patient eligibility criteria:

Inclusion criteria:

(i) Age ≥18 years; (ii) A new diagnosis of multiple myeloma or at progression of disease necessitating a change in treatment plan, or relapsed/refractory aggressive B cell lymphoma after one prior line of therapy; (iii) Eastern Cooperative Oncology Group (ECOG) performance status 0-3; (iv) Willingness to complete symptom screening; and (v) At least one ESAS-r-plus symptom scored at ≥3 at time of recruitment.

Exclusion criteria:

(i) Insufficient English literacy to complete study procedures; (ii) Hematologist-determined poor cognitive status; (iii) Current palliative care team involvement at PM or elsewhere; and (iv) Not receiving ongoing follow up with malignant hematology team at PM.

Caregiver eligibility criteria:

Inclusion criteria:

(i) Age ≥18 years; (ii) Caregiver of a patient with relapsed B cell lymphoma; and (iii) Willing to attend at least 1 PCC visit with the patient.

Exclusion criteria:

(i) Insufficient verbal and/or written English literacy to complete study procedures; or (ii) Patient not participating in study.

Healthcare provider eligibility criteria:

Inclusion criteria:

(i) Specialized staff physician, fellow, clinical nurse specialist, or clinic nurse from the outpatient malignant hematology team or palliative care team at PM working clinically with patients with multiple myeloma; and (ii) Working in their clinical area for at least 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of early palliative care for outpatients with multiple myeloma and aggressive lymphoma and their caregivers (lymphoma only) | 12 months
  The intervention will be feasible if the following criteria are met:
  (i) accrual of at least 80 patients (40 with multiple myeloma and 40 with aggressive B cell lymphoma) and up to 40 caregivers of patients with aggressive B cell lymphoma over 12 months; (ii) ≥60% of recruited patients and caregivers complete self-reported outcomes (PROs) at baseline, and monthly for three months; and (iii) ≥60% of patients and their caregivers in the intervention arm have at least one visit to the palliative care clinic.
Patient quality of life as measured by the FACIT-Pal | 3 months after enrollment
  The FACIT-Pal (Functional Assessment of Chronic Illness Therapy-Palliative Care) quality of life scale is a version of the 27-item FACT-G (Functional Assessment of Cancer Therapy-General) scale, with the addition of 19 items for patients with advanced illness. These 46 items measure physical, social/family, emotional, functional well-being, and additional concerns. Total scores range from 0-184, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Patient quality of life as measured by the FACIT-Pal | 1 month and 2 months after enrollment
  The FACIT-Pal (Functional Assessment of Chronic Illness Therapy-Palliative Care) quality of life scale is a version of the 27-item FACT-G (Functional Assessment of Cancer Therapy-General) scale, with the addition of 19 items for patients with advanced illness. These 46 items measure physical, social/family, emotional, functional well-being, and additional concerns. Total scores range from 0-184, with higher scores indicating better quality of life.
Patient symptom control as measured by the ESAS-r-CS | 1 month, 2 months, and 3 months after enrollment
  The ESAS-r-CS (Edmonton Symptom Assessment System-revised plus constipation and trouble sleeping) consists of 11 scales with anchors of 0 (best) and 10 (worst) with symptom descriptions for pain, fatigue, drowsiness, nausea, anxiety, depression, appetite, dyspnea, well-being. Individual symptom scores are summed for the ESAS Distress Score (9-items) and Total Distress Score (11-items). Individual scores range from 0-10, with lower scores indicating better symptom control.
Patient and caregiver depression as measured by the PHQ-9 | 1 month, 2 months, and 3 months after enrollment
  The PHQ-9 (Patient Health Questionnaire-9 item version) is a measure for screening, diagnosing, and monitoring the severity of depression. Total scores range from 0-27, with higher scores indicating worse depression.
Patient satisfaction with care as measured by the FAMCARE-P16 | 1 month, 2 months, and 3 months after enrollment
  The FAMCARE-P16 (FAMCARE satisfaction with care scale-16-item patient version) is a 16-item scale that measures patient satisfaction with information-giving, availability of care, psychological care and physical patient care in patients with advanced cancer. Total scores range from 16-80, with higher scores indicating greater satisfaction with care.
Patient performance status as measured by the PRFS | 1 month, 2 months, and 3 months after enrollment
  The PRFS (Patient-Reported Function Status) measures a patient's own activities and function on a five-point scale. It is based on the ECOG (Eastern Cooperative Oncology Group) performance scale, but is expressed in lay language. Total scores range from 0-4, with lower scores indicating better performance status.
Caregiver quality of life as measured by the CQOLC | 1 month, 2 months, and 3 months after enrollment
  The CQOLC (Caregiver Quality of Life Index-Cancer) is a 35-item measure of burden, disruptiveness, adaptation, financial, and additional caregiver concerns. Total scores range from 0-140, with higher scores indicating worse quality of life.
Caregiver satisfaction with patient care as measured by the FAMCARE-caregiver | 1 month, 2 months, and 3 months after enrollment
  The FAMCARE-caregiver is a 19-item caregiver version of the FAMCARE scale. Total scores range from 20-100, with higher scores indicating greater satisfaction with patient care.

CONTACTS AND LOCATIONS:
Overall Officials: Breffni Hannon, MB BCh BAO, MMedSci, MCFP, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No